CLINICAL TRIAL: NCT02714010
Title: Whole Brain Radiotherapy Concurrent With EGFR-TKI Versus EGFR-TKI Alone in the Treatment of Non-small Cell Lung Cancer Patients With Brain Metastasis
Brief Title: EGFR-TKI Concurrent With/Without WBRT in Brain Metastasis From NSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li-kun Chen, Associate Professor/Associate chief physician, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO1014
Record Dates: First submitted 2015-11-29; First posted 2016-03-21 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: EGFR-TKI; whole brain radiotherapy; brain metastasis; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Patients take EGFR-TKI alone till tumor progression
  Interventions: Drug: EGFR-TKI
- Arm 2 (Active Comparator): Patients take EGFR-TKI concurrent with whole brain radiotherapy (WBRT) till tumor progression, WBRT started within the first week of taking TKI
  Interventions: Drug: EGFR-TKI; Radiation: whole brain radiotherapy

INTERVENTIONS:
Drug: EGFR-TKI — Gefitinib 250mg po qd or Tarceva 150mg po qd or Icotinib 125mg po tid
  Other Names: Gefitinib/Tarceva/Icotinib
Radiation: whole brain radiotherapy — 30Gy/10F
  Other Names: WBRT
  Arms: Arm 2

SUMMARY:
This is a multi-center phase III randomized controlled study, designing to access whether the efficacy of EGFR-TKI alone on patients with brain metastasis from non-small cell lung cancer (NSCLC) harboring EGFR mutant type is not inferior to EGFR-TKI concurrent with whole brain radiotherapy (WBRT), the primary end point is intracranial PFS (iPFS), while secondary outcomes included overall survival (OS), objective response rate (ORR), evaluation of cognitive function, quality of life (QoL) and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients who was confirmed non-small cell lung cancer (NSCLC) by histology or cytology, harboring EGFR mutant type (19 and/or 21 exon mutation).
* Patients who was confirmed with asymptomatic, treatment naive brain metastasis (didn't receive any treatment after diagnosed with brain metastasis) by MRI, couldn't receive operation or stereotactic radiosurgery（SRS）.
* Appraisable disease, that is there must be at least one lesion with the longest diameter>10mm in brain (by brain MRI).
* Adult patients (18 to 75 years old). Eastern Cooperative Oncology Group（ECOG） performance status 0 to 2. Life expectancy of at least 12 weeks. Haemoglobin > 10g/dl, absolute neutrophil count (ANC) > 1.5 x 10^9/L, platelets > 100 x 10^9/L; total bilirubin < 1.5x upper limit of normal (ULN). Alanine aminotransferase（ALT） and aspartate aminotransferase（AST）< 1.5x ULN in the absence of liver metastases, or < 5x ULN in case of liver metastases. Creatinine clearance > 60ml/min (calculated according to Cockcroft-gault formula).
* Patients should be contraceptive during the period of the trial.

Exclusion Criteria:

* Patients who had received brain radiotherapy or EGFR-TKI before.
* Patients who can't receive WBRT.
* Uncontrolled intracranial hypertension after steroid or dehydration therapy.
* Patients who take phenytoin, Carbamazepine, Rifampicin, Barbital, or St John's Wort which will interfere with the metabolism of TKI.
* Patients with interstitial lung disease, significant ocular disease, or serious uncontrolled systematic disease.
* Patients who can't take oral tablets, with active peptic ulcer diseases.
* Pregnancy or breast-feeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Estimated)
Dates: Start 2015-08; Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
intracranial PFS (iPFS) | up to 41 months
  Compare intracranial PFS (iPFS) of two arms

SECONDARY OUTCOMES:
overall survival (OS) | up to 77 months
objective response rate (ORR) | up to 41 months

OTHER OUTCOMES:
cognitive impairment | up to 77 months
  questionnaire
quality of life (QoL) | up to 77 months
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: li-kun Chen, Principal Investigator — associate chief physician
Locations (1):
- Sun Yat-sen University of cancer center, Guangzhou, Guangdong, China